CLINICAL TRIAL: NCT05587309
Title: A Phase 3, Double-Blind, Randomized, Two-Phase, Active-Controlled Study to Evaluate the Efficacy and Safety of BLI5100 in Patients With Erosive Esophagitis
Brief Title: A Study to Evaluate the Efficacy and Safety of BLI5100 in Patients With Erosive Esophagitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Braintree Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BLI5100-301
Record Dates: First submitted 2022-10-17; First posted 2022-10-20 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Erosive Esophagitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Healing Phase - BLI5100 (Experimental): During the Healing Phase, patients will take BLI5100 once daily, orally, for up to 8 weeks.
  Interventions: Drug: BLI5100
- Healing Phase - PPI Control (Active Comparator): During the Healing Phase, patients will take a PPI control once daily, orally, for up to 8 weeks.
  Interventions: Drug: PPI Control
- Maintenance Phase - BLI5100 Low Dose (Experimental): During the Maintenance Phase, patients will take BLI5100 low dose once daily, orally, for 24 weeks.
  Interventions: Drug: BLI5100
- Maintenance Phase - BLI5100 High Dose (Experimental): During the Maintenance Phase, patients will take BLI5100 high dose once daily, orally, for 24 weeks.
  Interventions: Drug: BLI5100
- Maintenance Phase - PPI Control (Active Comparator): During the Maintenance Phase, patients will take a PPI control once daily, orally, for 24 weeks.
  Interventions: Drug: PPI Control

INTERVENTIONS:
Drug: BLI5100 — Orally via tablet
  Arms: Healing Phase - BLI5100; Maintenance Phase - BLI5100 High Dose; Maintenance Phase - BLI5100 Low Dose
Drug: PPI Control — Orally via tablet
  Arms: Healing Phase - PPI Control; Maintenance Phase - PPI Control

SUMMARY:
The objective of the Healing Phase of the study is to evaluate the safety and efficacy of up to 8 weeks of once daily oral administration of BLI5100 versus a PPI control in healing EE. The objective of the Maintenance Phase of the study is to evaluate the safety and efficacy of 24 weeks of once daily oral administration of BLI5100 (low or high dose) versus a PPI control in the maintenance of healed EE.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 years at the time of signing informed consent;
2. Have experienced both heartburn and regurgitation within 7 days prior to the Screening Visit;
3. Current evidence of EE of LA grades A to D based on an upper GI endoscopy;
4. Able to understand and comply with the protocol requirements;
5. Willing and able to provide written informed consent at Screening;
6. A female of reproductive potential defined as a non-post-menopausal female who has not had a bilateral oophorectomy or medically documented ovarian failure; or If a female of childbearing potential, agrees to use an acceptable form of birth control and avoid egg donation from the Screening Visit until 6 months after the last dose of study drug.
7. If a male, agrees to use an acceptable form of birth control from the Screening Visit until 3 months after the last dose of study drug.
8. If a male, agrees to abstain from sperm donation through 3 months after administration of the last dose of study drug.

Exclusion Criteria:

1. Unable to undergo an upper GI endoscopy;
2. Presence of esophageal stricture, gastroesophageal varix (including post sclerotherapy or ligation), untreated Barrett's esophagus, gastric bleeding, infection, tumor, or gastric or duodenal ulcer on the upper GI endoscopy;

   o Note: Patients with diagnosis of Schatzki's ring (mucosal tissue ring around lower esophageal sphincter) are eligible to participate.
3. Alarm symptoms such as odynophagia, severe dysphagia, upper GI bleeding, weight loss, anemia, or hematochezia within 4 weeks prior to Screening, unless the presumed malignancy is ruled out;
4. History of eosinophilic esophagitis, achalasia, or other primary esophageal motility disorder; functional heartburn; physiochemical trauma (including radiation, mucosal resection, or cryotherapy); or documented history of delayed gastric emptying;
5. History of a connective tissue disorder associated with GI symptoms (eg, scleroderma or systemic lupus erythematous) or inflammatory bowel disease;
6. History of acid-suppressive, esophageal, or gastric surgery;

   o Note: This is not applicable to appendectomy, cholecystectomy, or endoscopic excision of benign tumor.
7. History of malignancy within the past 5 years (with the exception of resected basal cell or squamous cell carcinoma of the skin);

   o Note: This is not applicable to patients who had complete response or pathological complete response and whose tumor had not recurred for at least 5 years from the date of last treatment, or patients whose tumor had been removed by endoscopic resection without any findings indicating recurrence of the tumor within 3 years.
8. History of an allergic disease, or hypersensitivity or intolerance to the active ingredient or excipients of the study drug;
9. History of alcoholism, chronic opiate use, or substance addiction in the 12 months before Screening or a positive urine drug screen for opiates or substances of abuse;

   * Note: Patients on prescribed opioids are eligible to participate if they have been on a stable dose for >3 months prior to Screening.
   * Note: Retesting of a positive urine drug screen requires Medical Monitor approval. Positive urine drug screen for all drugs will require verification of prescription for the positive tested substance.
10. Presence of manic-depression, anxiety disorder, panic disorder, somatoform disorder, personality disorder, or other psychological disorder;

    o Note: A diagnosis of manic-depression, anxiety disorder, panic disorder, somatoform disorder, personality disorder, or other psychological disorder is not exclusionary, as long as the patient is asymptomatic and well-controlled on stable treatment (ie, stable dose for >6 months prior to Screening), including non-medical therapy.
11. Current use of antipsychotics, antidepressants, anxiolytics, or prescription sleeping medications, with the exception of a stable dose for >6 months prior to Screening;
12. Use of any gastric acid-suppressive agents, including PPIs, within 2 weeks prior to the upper GI endoscopy at Screening;
13. Use of 2 or more commercial doses of ref lux esophagitis-related medications (including H2 blockers, prostaglandins, mucosal protective agents, and prokinetics) within 1 week prior to the upper GI endoscopy at Screening;
14. Requirement of persistent use of non-steroidal anti-inflammatory drugs (NSAIDs) during the course of the study;

    o Note: Low-dose (≤100 mg/day) aspirin is allowed provided that it has been used for prophylaxis prior to study participation.
15. If a female, is pregnant, breastfeeding, or planning to become pregnant during the study or within 6 months after the last dose of study drug;
16. Positive test result for human immunodeficiency virus, hepatitis B surface antigen, or hepatitis C virus at Screening;
17. Positive test result for H pylori at Screening or diagnosis and treatment of H pylori within 6 weeks prior to randomization;

    o Note: Patients who test positive for H pylori at Screening will be offered treatment according to local standard of care and may be re-screened for eligibility following completion of treatment.
18. Abnormal laboratory results with clinical relevance at Screening as follows:

    * Aspartate aminotransferase (AST), ALT, or alkaline phosphatase level of ≥2 × upper limit of normal (ULN);
    * Total bilirubin level of ≥2 × ULN, unless Gilbert's syndrome is confirmed when direct bilirubin is ≤0.3 mg/dL;
    * Estimated glomerular filtration rate <30 mL/min; or
    * Serum magnesium < lower limit of normal.
19. Abnormal ECG of clinical significance (eg, major arrhythmia, multifocal premature ventricular contractions, or 2° atrioventricular block anomaly);
20. Presence of any gastric acid hypersecretory conditions, such as Zollinger-Ellison syndrome;
21. Involvement in another clinical study within 4 weeks of initiation of study drug;
22. Any other clinically relevant condition that would confound study endpoints or adversely affect patient compliance with the study procedures in the medical judgment of the Investigator or Medical Monitor based on previous medical history or findings on Screening assessments.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1250 (Actual)
Dates: Start 2022-10-30 (Actual); Primary Completion 2025-06-16 (Actual); Study Completion 2025-06-16 (Actual)

PRIMARY OUTCOMES:
Healing Phase: Percentage of patients with complete healing by Week 8. | 8 Weeks
Maintenance Phase: Percentage of patients who maintain complete healing through Week 24. | 24 Weeks

SECONDARY OUTCOMES:
Healing Phase: Percentage of 24-hour heartburn-free days through Week 8. | 8 Weeks
Maintenance Phase: Percentage of 24-hour heartburn-free days through Week 24. | 24 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Leah Hollins, Study Director — Braintree Laboratories / Sebela Pharmaceuticals
Locations (122):
- United States (122):
  - Research Site 145, Homewood, Alabama
  - Research Site 24, Huntsville, Alabama
  - Research Site 132, Peoria, Arizona
  - Research Site 150, Peoria, Arizona
  - Research Site 62, Phoenix, Arizona
  - Research Site 27, Tucson, Arizona
  - Research Site 87, Little Rock, Arkansas
  - Research Site 117, North Little Rock, Arkansas
  - Research Site 51, Arcadia, California
  - Research Site 66, Bell Gardens, California
  - Research Site 156, Camarillo, California
  - Research Site 19, Canoga Park, California
  - Research Site 94, Chula Vista, California
  - Research Site 10, Huntington Park, California
  - Research Site 55, La Mesa, California
  - Research Site 72, Los Angeles, California
  - Research Site 14, San Diego, California
  - Research Site 85, Santa Ana, California
  - Research Site 13, Santa Ana, California
  - Research Site 41, Santa Maria, California
  - Research Site 54, Westlake, California
  - Research Site 89, Littleton, Colorado
  - Research Site 147, Bristol, Connecticut
  - Research Site 74, Boca Raton, Florida
  - Research Site 108, Cooper City, Florida
  - Research Site 91, Doral, Florida
  - Research Site 03, Hialeah, Florida
  - Research Site 78, Homestead, Florida
  - Research Site 09, Lake City, Florida
  - Research Site 23, Maitland, Florida
  - Research Site 38, Miami, Florida
  - Research Site 43, Miami, Florida
  - Research Site 67, Miami, Florida
  - Research Site 92, Miami, Florida
  - Research Site 31, Miami, Florida
  - Research Site 71, Miami, Florida
  - Research Site 42, Miami Lakes, Florida
  - Research Site 17, New Port Richey, Florida
  - Research Site 90, Ocoee, Florida
  - Research Site 107, Orlando, Florida
  - Research Site 05, Palmetto Bay, Florida
  - Research Site 95, St. Petersburg, Florida
  - Research Site 11, Sunrise, Florida
  - Research Site 46, Viera, Florida
  - Research Site 153, Atlanta, Georgia
  - Research Site 04, Marietta, Georgia
  - Research Site 59, Sandy Springs, Georgia
  - Research Site 151, Boise, Idaho
  - Research Site 101, Idaho Falls, Idaho
  - Research Site 143, Glenview, Illinois
  - Research Site 01, Gurnee, Illinois
  - Research Site 141, Gurnee, Illinois
  - Research Site 02, Oak Lawn, Illinois
  - Research Site 135, South Bend, Indiana
  - Research Site 125, Covington, Louisiana
  - Research Site 45, Houma, Louisiana
  - Research Site 12, Marrero, Louisiana
  - Research Site 124, Metairie, Louisiana
  - Research Site 48, Metairie, Louisiana
  - Research Site 34, New Orleans, Louisiana
  - Research Site 25, West Monroe, Louisiana
  - Research Site 93, Chesterfield, Michigan
  - Research Site 148, Plymouth, Minnesota
  - Research Site 140, Flowood, Mississippi
  - Research Site 111, Chesterfield, Missouri
  - Research Site 137, Columbia, Missouri
  - Research Site 138, Kansas City, Missouri
  - Research Site 159, Henderson, Nevada
  - Research Site 160, Las Vegas, Nevada
  - Research Site 73, Las Vegas, Nevada
  - Research Site 06, Las Vegas, Nevada
  - Research Site 163, Las Vegas, Nevada
  - Research Site 127, Las Vegas, Nevada
  - Research Site 64, Reno, Nevada
  - Research Site 129, Englewood, New Jersey
  - Research Site 130, Freehold, New Jersey
  - Research Site 131, Jackson, New Jersey
  - Research Site 35, Brooklyn, New York
  - Research Site 07, Great Neck, New York
  - Research Site 28, Hartsdale, New York
  - Research Site 58, New York, New York
  - Research Site 49, New York, New York
  - Research Site 40, Rochester, New York
  - Research Site 75, Fayetteville, North Carolina
  - Research Site 155, High Point, North Carolina
  - Research Site 69, Mount Airy, North Carolina
  - Research Site 116, Salisbury, North Carolina
  - Research Site 158, Columbus, Ohio
  - Research Site 20, Columbus, Ohio
  - Research Site 88, Columbus, Ohio
  - Research Site 109, Mentor, Ohio
  - Research Site 118, Springboro, Ohio
  - Research Site 110, Westlake, Ohio
  - Research Site 157, Anderson, South Carolina
  - Research Site 61, North Charleston, South Carolina
  - Research Site 128, Hermitage, Tennessee
  - Research Site 114, Kingsport, Tennessee
  - Research Site 60, Nashville, Tennessee
  - Research Site 103, Nashville, Tennessee
  - Research Site 50, Shelbyville, Tennessee
  - Research Site 100, Bellaire, Texas
  - Research Site 98, Dallas, Texas
  - Research Site 99, Forney, Texas
  - Research Site 154, Houston, Texas
  - Research Site 162, Houston, Texas
  - Research Site 68, Katy, Texas
  - Research Site 29, Lewisville, Texas
  - Research Site 161, McAllen, Texas
  - Research Site 32, Pearland, Texas
  - Research Site 30, Red Oak, Texas
  - Research Site 22, San Antonio, Texas
  - Research Site 26, San Antonio, Texas
  - Research Site 21, San Antonio, Texas
  - Research Site 80, Tomball, Texas
  - Research Site 134, Waco, Texas
  - Research Site 105, Ogden, Utah
  - Research Site 57, Salt Lake City, Utah
  - Research Site 65, Sandy City, Utah
  - Research Site 16, South Ogden, Utah
  - Research Site 77, Chesapeake, Virginia
  - Research Site 136, Richmond, Virginia
  - Research Site 97, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No